CLINICAL TRIAL: NCT05867017
Title: Long-Term Sequelae of SARS-COV-2 Infection: Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HSC20220656H; OT2HL161847-01 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-05-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: COVID-19; Diabete Mellitus
Keywords: Glycemic control; Long term medical effects of COVID-19; Blood glucose control; Insulin sensitivity
MeSH Terms: conditions — COVID-19; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Plasma samples for future lipidomic and metabolomic analysis will be frozen at -80degC for later analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe COVID-19 Group: Hospitalized in ICU with COVID-19 (PCR positive) and recovered
  Interventions: Other: Measure of physiologic parameters
- Mild COVID-19 positive Group: COVID-19 positive (by PCR) who recovered from mild COVID-19 and were seen in outpatient clinics or ER with symptoms that did not justify hospitalization.
  Interventions: Other: Measure of physiologic parameters
- COVID-19 negative Group: COVID-19 negative (by PCR) and seen in outpatient clinics or ER during same time period as Groups I and II.
  Interventions: Other: Measure of physiologic parameters

INTERVENTIONS:
Other: Measure of physiologic parameters — Participants will have hepatic muscle and adipose tissue insulin sensitivity tested

SUMMARY:
Hospitalized patients with severe COVID-19 have an increased incidence of insulin resistance, impaired beta cell function, glucose intolerance (prediabetes), and overt type 2 diabetes (T2D) compared to non-hospitalized patients with COVID-19 and COVID-19 negative individuals on long-term follow up.

DETAILED DESCRIPTION:
The purpose of this research study is to understand the long-term effects of COVID-19 infection on individuals without any prior history of diabetes. This study will look at several measures of diabetes, such as glycemic control (blood glucose/sugar levels), function of beta cells (cells that make insulin to control sugar), insulin secretion and insulin sensitivity (fasting insulin levels).

The following participants will be enrolled: 1) have had COVID-19 infection and were hospitalized and recovered, or 2) have had mild COVID-19 infection and were seen at outpatient clinics or ER and were not required to be hospitalized, or 3) have not had COVID-19 infection but were seen in outpatient clinics or ER during the same time period.

The researchers hope to learn the long-term effects of COVID-19 infection in hospitalized patients. Specifically, they will be focusing on the subsequent development of diabetes and associated metabolic disturbances, such as impaired insulin secretion and insulin resistance. A relationship between COVID-19 and diabetes needs to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index (BMI) < 40 kg/m2

Exclusion Criteria:

* History of diabetes prior to SARS-CoV-2 infection
* Took medications used to treat diabetes prior to SARS-CoV-2 infection
* History of myocardial infarction or stroke within 6 months
* History of major organ system disease prior to COVID-19 infection

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Three groups from background (general) population including Mexican ancestry will be studied, who have no history of diabetes or treatment with diabetes drugs prior to COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Measure of glycosylated glucose percentage (HbA1c) | Baseline to 24 months
  Change in HbA1c, and indication of glucose levels over a 3 month period
Measure of free plasma glucose (FPG) | Baseline to 24 months
  Change in FPG

SECONDARY OUTCOMES:
Body Weight | Baseline to 24 months
  Change in body weight over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Texas Diabetes Institute - University Health System, San Antonio, Texas, United States